CLINICAL TRIAL: NCT02079220
Title: A Phase II Study of Ziv-aflibercept in Combination With Capecitabine/Oxaliplatin (XELOX) Chemotherapy in the Front-Line Treatment of Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding for the study was withdrawn, no participants were ever recruited.
Sponsor: James J Lee (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, James J Lee, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-145
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal Cancer; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Arm A (every 2 week schedule) Dosage and dosage regimen for all study periods
  * Capecitabine: will be administered 1,000 mg/m2 orally twice a day on Days 1 - 7 of each cycle, repeating every 14 days.
  * Oxaliplatin: will be administered 85 mg/m2 IV on Day 1 of each cycle, repeating every 14 days.
  * Ziv-aflibercept: will be administered 4 mg/kg IV on Day 1 of each cycle, repeating every 14 days.
  Interventions: Drug: Arm A
- Arm B (Experimental): Arm B (every 3 week schedule):
  Dosage and dosage regimen for all study periods
  * Capecitabine: will be administered 850 mg/m2 orally twice a day on Days 1 - 14 of each cycle, repeating every 21 days.
  * Oxaliplatin: will be administered 130 mg/m2 IV on Day 1 of each cycle, repeating every 21 days.
  * Ziv-aflibercept: will be administered 6 mg/kg IV on Day 1 of each cycle, repeating every 21 days.
  Interventions: Drug: Arm B

INTERVENTIONS:
Drug: Arm A — * Capecitabine
  * Oxaliplatin
  * Ziv-aflibercept
  Other Names: Xeloda; ELOXATIN; ZALTRAP
  Arms: Arm A
Drug: Arm B — Capecitabine Oxaliplatin Ziv-aflibercept
  Other Names: Xeloda; ELOXATIN; ZALTRAP
  Arms: Arm B

SUMMARY:
This is an open label, two-arm, phase II trial to evaluate the anti-tumor activity, safety, and tolerability of ziv-aflibercept in combination with XELOX chemotherapy in the first-line treatment of subjects with mCRC.

Two different schedules of ziv-aflibercept in combination with XELOX will be evaluated in this study: every 2 week schedule (Arm A) and the every 3 week schedule (Arm B). The choice between arm A and arm B will depend on the investigator's preference.

Arm A (every 2 week schedule) Dosage and dosage regimen for all study periods

* Capecitabine: will be administered 1,000 mg/m2 orally twice a day on Days 1 - 7 of each cycle, repeating every 14 days.
* Oxaliplatin: will be administered 85 mg/m2 IV on Day 1 of each cycle, repeating every 14 days.
* Ziv-aflibercept: will be administered 4 mg/kg IV on Day 1 of each cycle, repeating every 14 days.

Arm B (every 3 week schedule):

Dosage and dosage regimen for all study periods

* Capecitabine: will be administered 850 mg/m2 orally twice a day on Days 1 - 14 of each cycle, repeating every 21 days.
* Oxaliplatin: will be administered 130 mg/m2 IV on Day 1 of each cycle, repeating every 21 days.
* Ziv-aflibercept: will be administered 6 mg/kg IV on Day 1 of each cycle, repeating every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* The study will be limited to subjects with newly diagnosed mCRC without any prior systemic chemotherapy for metastatic disease.
* The diagnosis of metastatic colorectal cancer will be based on histologic or cytologic confirmation.
* Subjects must have the ability to swallow oral medication.
* Subjects must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Any prior chemotherapy for mCRC is not allowed. Adjuvant chemotherapy with oxaliplatin-containing regimen CRC within the last 12 months is not allowed. Adjuvant chemotherapy with Fluorouracil (5-FU) or capecitabine alone within the last 6 months is allowed.
* Age ≥ 18 years.
* Both men and women of all races and ethnic groups are eligible for this trial.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (Karnofsky ≥ 60%).
* Life expectancy of greater than 12 months.
* Patients must have normal organ and marrow function as defined below:

  * Absolute Neutrophil Count ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Total Bilirubin 2 × institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and Alanine transaminase (ALT) 2.5 × institutional upper limit of normal (AST and ALT ≤ 5.0 x ULN is acceptable if liver has tumor involvement).
  * Creatinine Clearance (CrCl) 30 mL/min.
* The effects of the combination of ziv-aflibercept, oxaliplatin and capecitabine on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and 6 months after last administration of ziv-aflibercept. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of therapeutic agents administration and 6 months after last administration of ziv-aflibercept.
* Ability to understand and to sign a written informed consent document.

Exclusion Criteria:

* Unwilling or unable to follow protocol requirements or to give informed consent.
* Any prior chemotherapy for mCRC.
* Adjuvant chemotherapy with oxaliplatin-containing regimen CRC within the last 12 months.
* Adjuvant chemotherapy with 5-FU or capecitabine alone within the last 6 months is allowed.
* CrCl < 30 mL/min
* Any peripheral neuropathy of grade ≥ 2
* Patients with known dihydropyrimidine dehydrogenase (DPD) deficiency
* Patients with urine protein creatinine ration > 1 or urine protein > 500 mg/24 hours.
* Patients who have had radiotherapy within 4 weeks to entering the study or those who have not recovered from adverse events due to radiotherapy administered more than 4 weeks earlier.
* Patients with uncontrolled or symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Presence of metastatic disease that, in the opinion of the investigator, would require palliative treatment within 4 weeks of enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ziv-aflibercept, capecitabine, and oxaliplatin are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ziv-aflibercept, capecitabine, and oxaliplatin, breastfeeding should be discontinued if the mother is treated with ziv-aflibercept, capecitabine, and oxaliplatin.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ziv-aflibercept, capecitabine, and oxaliplatin. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.
* Serious or non-healing wound, skin ulcer, or bone fracture.
* History of bleeding diathesis or coagulopathy or active anticoagulation with Coumadin.
* Any documented stroke or Transient Ischemic Attack (TIA) within 6 months prior to study entry
* Any grade 3/4 hemorrhage within 3 months prior to study entry
* Any pulmonary embolism (PE) within 3 months prior to study entry
* Any deep vein thrombosis (DVT) within 3 months prior to study entry
* Uncontrolled hypertension defined as > 140/90 mmHg or isolated systolic hypertension > 160 mmHg on 2 separate days in past 3 months prior to study inclusion.
* Any of the following cardiac conditions:

  * Documented congestive heart failure
  * Myocardial infarction within 6 months prior to study entry
  * Unstable angina within 6 months prior to study entry
  * Symptomatic arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
anti-tumor activity of ziv-aflibercept in combination with XELOX in the first-line treatment of patients with metastatic colorectal cancer (mCRC) | up to 6 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States